CLINICAL TRIAL: NCT02114242
Title: Development of Biomarkers for the Diagnosis and Prognosis of Parkinsonian Syndromes Running Head: Biomarkers in Parkinsonian Syndromes
Brief Title: Biomarkers in Parkinsonian Syndromes
Acronym: BIOPARK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2012/27
Record Dates: First submitted 2014-02-06; First posted 2014-04-15 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Parkinsonian Syndromes; Parkinson's Disease; Multiple System Atrophy; Progressive Supranuclear Palsy
Keywords: Parkinson's disease; multiple system atrophy; progressive supranuclear palsy; alpha-synuclein
MeSH Terms: conditions — Parkinsonian Disorders; Parkinson Disease; Multiple System Atrophy; Supranuclear Palsy, Progressive; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Cerebrospinal fluid
  * Whole blood
  * Plasma
  * Serum
  * Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Parkinson's disease patients: Patients suffering from Parkinson desease
  Interventions: Other: clinical measures of disease severity and progression
- multiple system atrophy patients: Patients suffering from "probable" multiple system atrophy according to clinical consensus criteria and age > 30
  Interventions: Other: CSF, blood and urine sampling; Other: clinical measures of disease severity and progression
- progressive supranuclear palsy: Patients suffering from progressive supranuclear palsy and age > 40
  Interventions: Other: CSF, blood and urine sampling; Other: clinical measures of disease severity and progression

INTERVENTIONS:
Other: CSF, blood and urine sampling — PSP and MSA patients will receive CSF and blood sampling at two study visits (baseline and after 12 months).
  Groups: multiple system atrophy patients; progressive supranuclear palsy
Other: clinical measures of disease severity and progression — Questionnaires (quality of life, motricity scales, cognitive scales, depression scales, scale of sleep quality)

SUMMARY:
Parkinson disease (PD), multiple system atrophy (MSA) and progressive supranuclear palsy (PSP) are neurodegenerative disorders. PD and MSA are alpha-synucleinopathies, which are characterized by the abnormal accumulation of alpha-synuclein, while tau protein accumulates in PSP. The development of biological markers for the diagnosis and prognosis in PD, MSA and PSP remains an unmet need. Such biological markers are crucial for future disease-modification and neuroprotection trials. Alpha-synuclein has a high potential for biomarker development since it constitutes the pathological hallmark feature in PD and MSA. The oligomeric alpha-synuclein seems to be particularly involved in abnormal protein aggregation in alpha-synucleinopathies.

The main objective is to compare oligomeric alpha-synuclein CSF levels between PD, MSA and PSP patients. PD and MSA patients will receive Cerebrospinal Fluid (CSF) and blood sampling at two study visits (baseline and after 12 months). Major secondary objectives are (i) to assess potential associations between the biomarker and clinical measures of disease severity and progression in MSA and PSP, and (ii) to assess the variation of the biomarker and its correlation to disease severity and progression in PD, MSA and PSP.

DETAILED DESCRIPTION:
The differential diagnosis between Parkinson's disease, multiple system atrophy and progressive supranuclear palsy can be very difficult in early disease. PD, MSA and PSP are neurodegenerative disorders. PD and MSA belong to the alpha-synucleinopathies, which are characterized by the abnormal accumulation of alpha-synuclein. Alpha-synuclein accumulates in intraneuronal Lewy bodies in PD patients and as intracytoplasmic glial inclusions in MSA. In PSP, tau protein accumulates in neurons and glia cells while alpha-synuclein deposits are only found to a small extend.

The development of biological markers for the diagnosis and prognosis of PD, MSA and PSP remains an unmet need. Beyond guiding clinical decision-making, such biological markers are crucial for future disease-modification and neuroprotection trials.

Alpha-synuclein has a high potential for biomarker development since it constitutes the pathological hallmark feature of PD and MSA. The oligomeric alpha-synuclein fraction whose CSF levels are increased in PD seems to be particularly involved in abnormal protein aggregation in alpha-synucleinopathies.

The main objective of the study is to compare oligomeric alpha-synuclein CSF levels between PD, MSA and PSP patients. Secondary objectives are (i) to compare total alpha-synuclein levels and the index total/oligomeric alpha-synuclein between PD, MSA and PSP, (ii) to study the correlation and concordance between CSF and plasma levels of total and oligomeric alpha-synuclein, (iii) to assess potential associations between the biomarker and clinical measures of disease severity and progression and (iv) to assess the variation of the biomarker over time and its correlation to disease severity and progression.

ELIGIBILITY:
Patients receiving anticoagulants, showing abnormal coagulation on blood testing or thrombocytopenia are excluded from this study.

Patients showing more than 500 erythrocytes per mm3 of LCR are excluded from this study.

* PD patients

  * inclusion criteria:

    * Patients suffering from PD according to clinical criteria (Hughes et al, 1992)
    * Written informed consent
    * Patient covered by the national health system
  * exclusion criteria:

    * Patient under tutelage
    * patient covered by the national health system
* MSA patients

  * inclusion criteria:

    * Patients suffering from "possible" or "probable" MSA according to clinical consensus criteria (Gilman et al, 2008), age > 30
    * Written informed consent
    * Patient covered by the national health system
  * exclusion criteria:

    * UMSARS IV score >4 points
    * Patient under tutelage
* PSP patients

  * inclusion criteria:

    * Patients suffering from PSP according to NNIPPS trial criteria (Bensimon et al., 2009), age > 40
    * Written informed consent
    * Patient covered by the national health system
  * exclusion criteria:

    * PSPRS item 26 score >3 points
    * Patient under tutelage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from parkinson disease or multiple system atrophy or progressive supranuclear palsy.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-12-16 (Actual); Primary Completion 2023-12-16 (Estimated); Study Completion 2025-12-16 (Estimated)

PRIMARY OUTCOMES:
Concentration of oligomeric alpha-synuclein in cerebrospinal fluid | at day 0 (inclusion) and one year after inclusion

SECONDARY OUTCOMES:
Total alpha-synuclein concentration in CSF, oligomeric/total alpha-synuclein ratio in CSF | At inclusion (Day 0) and one year after inclusion
Oligomeric and total alpha-synuclein concentration in plasma, oligomeric/total alpha-synuclein ratio in plasma | At inclusion (Day 0) and one year after inclusion
Alpha-synuclein levels in relation to disease severity and progression, disease duration and age | At inclusion (Day 0) and one year after inclusion
Variation of alpha-synuclein levels between first and second sampling | At inclusion (Day 0) and one year after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Wassilios MEISSNER, Pr, Principal Investigator — University Hospital, Bordeaux; Rodolphe THIEBAUT, MD, Study Chair — University Hospital, Bordeaux
Locations (3):
- France (3):
  - CHU de Limoges, Limoges
  - CHU de Bordeaux, Pessac
  - CHU de Toulouse, Toulouse